CLINICAL TRIAL: NCT02743975
Title: Intraoperative Detection of Cancer Tissue in Pancreatic Adenocarcinoma Using a VEGF-targeted Optical Fluorescent Imaging Tracer, A Multicentre Feasibility Dose Escalation Study
Brief Title: Near-infrared Image Guided Surgery in Pancreatic Adenocarcinoma
Acronym: PENGUIN
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Insufficient tumor-to-background ratios in the first three dose groups
Sponsor: University Medical Center Groningen (Other)
Collaborators: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, G.M. van Dam, Prof. Dr., University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL50488.042.15
Record Dates: First submitted 2016-04-11; First posted 2016-04-19 (Estimated); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Pancreatic Cancer; Pancreatic Adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: phase I/II safety and dose-finding study
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment group (Experimental): Bevacizumab-800CW
  Interventions: Drug: Bevacizumab-800CW

INTERVENTIONS:
Drug: Bevacizumab-800CW — dose finding: 4.5mg; 10mg; 25mg; 50mg
  Other Names: Bevacizumab-IRDye800CW

SUMMARY:
There is a need for better visualization of resection margins and detection of small tumor deposits during surgery for pancreatic cancer. Optical molecular imaging of pancreatic ductal adenocarcinoma associated biomarkers is a promising technique to accommodate this need. The biomarker Vascular Endothelial Growth Factor (VEGF-A) is overexpressed in pancreatic cancer tissue versus normal tissue and has proven to be a valid target for molecular imaging. VEGF-A can be targeted by the monoclonal antibody bevacizumab. Monoclonal antibodies can be labeled by the near-infrared (NIR) fluorescent dye IRDye800CW (800CW). The investigators hypothesize that bevacizumab-800CW accumulates in VEGF expressing cancer, enabling pancreatic cancer visualization using a NIR intraoperative camera system. In this pilot intervention study the investigators will determine the optimal dosage of bevacizumab-800CW (4,5 10, 25 or 50mg) to detect pancreatic cancer tissue intraoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Patients with clinical suspicion of pancreatic head cancer who are scheduled to undergo surgical intervention with curative intent
* World Health Organization (WHO) performance score 0-2.
* Signed written informed consent

Exclusion Criteria:

* Medical or psychiatric conditions that compromise the patient's ability to give informed consent.
* Other invasive malignancy
* Pregnant or lactating women. Documentation of a negative pregnancy test must be available for woman of childbearing potential. Woman of childbearing potential are pre- menopausal women with intact reproductive organs and women less than two years after menopause.
* Prior neo-adjuvant chemo- of radiotherapy
* History of infusion reactions to bevacizumab or other monoclonal antibody therapies.
* Inadequately controlled hypertension with or without current antihypertensive medications
* Within 6 months prior to inclusion: myocardial infarction, Transient Ischemic Attack, Cerebral Vascular Accident, pulmonary embolism, uncontrolled chronic hepatic failure, unstable angina pectoris.
* Anticoagulant therapy with vitamine K antagonists
* Patients receiving Class 1A (quinidine, procainamide) or class III (dofetilide, amiodarone, sotalol) antiarrhythmic agents
* Evidence of QTc (corrected QT interval) prolongation on pretreatment ECG (greater than 44ms in males of greater than 450ms in females)
* Magnesium, potassium and calcium below the lower limit of normal range.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-02-26 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Tracer accumulation in tumor tissue vs normal pancreatic tissue assessed by intraoperatively and ex vivo measuring of the mean fluorescent intensity | up to 6 months
  Mean Fluorescent Intensity (MFI) measured in tumor tissue compared to normal pancreatic tissue at macroscopic and microscopic level
Finding optimal dose of Bevacizumab-800CW for intraoperative imaging of pancreatic cancer measured by calculating Target to Background ratios (TBR) | 3 days after tracer injection
  TBR of each dose group assessed by intraoperative imaging as well as ex vivo imaging

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events | Up to 4 weeks after tracer injection

CONTACTS AND LOCATIONS:
Overall Officials: Gooitzen van Dam, MD, Principal Investigator — University Medical Center Groningen
Locations (3):
- Netherlands (3):
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Center, Leiden
  - Radboud University Medical Center, Nijmegen

IPD SHARING:
Plan to Share IPD: Undecided